CLINICAL TRIAL: NCT03658226
Title: A Case Series Evaluation of Psychodynamic Interpersonal Therapy (PIT) in Chronic Low Back Pain (CLBP) Patients
Brief Title: Case Series Evaluation of Psychodynamic Interpersonal Therapy in Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charlotte Morgan (Other)
Responsible Party: Sponsor-Investigator, Charlotte Morgan, Trainee Clinical Psychologist, University of Manchester
Organization: University of Manchester (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NHS001382
Record Dates: First submitted 2018-05-23; First posted 2018-09-05 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Chronic Low Back Pain
Keywords: Case Series; Acceptability; Feasibility; Psychodynamic Interpersonal Therapy

STUDY DESIGN:
Intervention Model Description: A series of experimental single case studies comparing individual CLBP participants' clinical outcomes during a baseline phase (receive no treatment) with those during a treatment phase (receive 8 sessions of PIT). Clinical outcomes will be the impact of treatment on pain distress/intensity, self-efficacy, mood and interpersonal functioning. There will be repeated measurement (daily/weekly) of the outcomes during baseline and intervention phases, to assess real-time change in these variables on a case-by-case basis. We will vary the length of the baseline phase randomly across participants, who will commence treatment following 3, 4, 5 or 6 weeks. This "multiple baselines" design will allow us to establish whether any improvement in clinical outcomes is caused by the intervention rather than natural change over time. We will assess feasibility/acceptability of the intervention by recording adverse reactions, side effects, adherence and participants' views about the intervention.
Masking Description: The PI/therapist will be blind to the outcome measures. All measures will be marked with a participant ID by an alternative researcher so that the therapist/PI will be unaware of individual participants' scores when analysing the data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therapy (Experimental): Psychodynamic Interpersonal Therapy (PIT)
  Interventions: Behavioral: Psychodynamic Interpersonal Therapy (PIT)

INTERVENTIONS:
Behavioral: Psychodynamic Interpersonal Therapy (PIT) — PIT is conversational model of psychotherapy; participants will receive 8 sessions of this therapy once weekly. The first session will be 2 hours and all remaining sessions will be 50 minutes.

SUMMARY:
Many people in the world have chronic pain; this is pain which lasts more than twelve weeks. Pain can cause people to feel low in mood and change how they feel about themselves and others around them. Therapy for chronic pain does not always work and often people do not have lasting effects from treatment. This study hopes to see if a different therapy, called Psychodynamic Interpersonal Therapy (PIT), can help people with chronic pain. This therapy looks at how we see ourselves and our relationships with others; it aims to help people address personal problems that make it difficult for them to manage their pain.

The study aims to show that PIT is a suitable treatment for chronic low back pain and that people will have fewer problems with their mood, how they feel about themselves and their relationships. This study will give people with chronic low back pain eight sessions of PIT and during therapy they will fill in forms about their pain, mood, relationship problems and how they feel about themselves. We will also look at practical things to do with the therapy (e.g. how many sessions people came to, reasons for stopping therapy etc.) and ask people about how they felt about the therapy they had. Three months after the study has finished, people will be asked to fill in the forms again to see if the effects have lasted.

This research could help to give people with chronic pain a new and different treatment option which has good and lasting effects.

DETAILED DESCRIPTION:
Chronic pain is continuous, long-term pain of more than 12 weeks. Patients with chronic pain are a heterogeneous group with varied pathologies (e.g. osteoarthritis; fibromyalgia) and pain sites (e.g., chronic low back pain, CLBP; chronic widespread pain). Chronic pain affects more than two fifths of the UK population, that is, around 28 million adults. Currently, the biopsychosocial model of pain is the most widely used heuristic approach to understanding chronic pain. The biopsychosocial perspective recognises that pain emerges from a dynamic interplay of a patient's physiological state, thoughts, emotions, behaviours, and sociocultural influences. This acknowledges that pain is a subjective experience and treatment approaches are aimed at management, rather than cure, of chronic pain.

Chronic pain affects social, psychological and emotional wellbeing. Current psychological treatments (e.g. CBT and ACT) aim to support patients to cope with the impact of chronic pain and improve their quality of life. However, some critical questions remain regarding the effectiveness of these interventions. Research indicates that substantial numbers of patients do not benefit greatly from these approaches and often effects are not maintained across time. Audit data from a local Pain Management Programme (PMP) indicates that many patients remain distressed by pain after treatment, with approximately 80% scoring 5 or more out of 10 on a pain distress scale six months later. Thus, it appears that current psychological therapies are not targeting all relevant issues.

Evidence indicates that psychodynamic therapies show some efficacy in the treatment of chronic pain, demonstrating patterns of change in interpersonal problems, pain intensity and depression-anxiety. Interpersonal literature states that aspects of relating are implicated in chronic pain; for example, perceived burdensomeness (feeling a burden on others) and thwarted belongingness (loneliness and feeling alienated from others) are significantly associated with pain intensity, self-efficacy and functional limitations.

Psychodynamic Interpersonal Therapy affirms that our sense of self and ability to relate to others are important determinants of how able we are to regulate emotion, manage adversity and access social support. As such, they are likely to play a fundamental role in how we cope with chronic pain. Studies have found an association between insecure attachment and related interpersonal difficulties with poor pain self-efficacy, anxiety and poor coping. Therefore, a psychological therapy such as PIT which focuses on addressing negative relationship patterns and strengthening sense of self may be of value in the treatment of chronic pain.

Psychological interventions such as PMPs seek to address the role of relationships and social networks in self-management of pain but do not target the psychological issues underlying interpersonal problems. Where individuals report high levels of interpersonal difficulties, a more in-depth focus on these issues may be required. As PIT seeks to understand how problematic patterns of relating are contributing to a person's distress and maladaptive coping, it may be a helpful approach. A clinical example of this is a person whose pain is exacerbated by overactivity related to their inability to say no to other's demands (e.g. for fear of upsetting them or eliciting conflict and rejection). Additionally, PIT has many strengths as an approach; it is a short, manualised and evidence-based treatment which has previously demonstrated promising results in the treatment of other conditions characterised by disabling chronic pain such as multisomatoform functional syndromes disorder and irritable bowel syndrome.

Presently, the efficacy of PIT in chronic pain is unknown. With that in mind, the proposed study seeks to conduct an evaluation of the acceptability, feasibility and efficacy of PIT in a chronic pain population; treatment resistant CLBP. The outcome of this study has the potential to inform future therapeutic options for those with chronic pain. The results may support the use of an alternative 1:1 therapy for those with interpersonal difficulties as it follows that they would require a treatment for chronic pain which has an interpersonal focus.

The primary aim of this study is to conduct a preliminary evaluation of whether PIT is an acceptable and feasible therapy for patients with treatment resistant CLBP (where patients are still experiencing clinically significant pain following previous treatment) and interpersonal difficulties. This will be measured using adherence to therapy and patient satisfaction and acceptability measures.

The secondary aim is to conduct an initial evaluation of the efficacy of PIT in people with treatment resistant CLBP and interpersonal problems, including its impact on pain distress, self -efficacy, and interpersonal functioning.

ELIGIBILITY:
Inclusion Criteria:

* Previously attended the Walton Centre pain management programme (PMP).
* Treatment resistant; six months after PMP treatment still experiencing clinically significant pain measured as 5+ on the pain distress rating scale. IMMPACT recommendations advise the use of numerical rating scales (NRS) in clinical trials of chronic pain treatments (Dworkin et al., 2005).
* Classified as "interpersonally distressed" on the West Haven Yale Multidimensional Pain Inventory (WHYMPI).
* Able to converse in English proficiently which is a requirement given the conversational nature of therapy.
* Able to commit to treatment and willing to be randomly allocated to baseline.

Exclusion Criteria:

* Other comorbid degenerative conditions and cancers.
* Psychosis
* History of prior suicide attempts.
* Active plans of self-harm and/or suicide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-09-09 (Actual)

PRIMARY OUTCOMES:
Objective measure of behaviour 1 - Number of sessions attended | Measured at the end of therapy (at week 8).
  Measuring feasibility/acceptability of therapy
Satisfaction questionnaire (PIT for CLBP) | Administered twice in the 8 weeks of therapy after session 1 (week 1) and Session 8 (week 8); the first and last sessions of therapy.
  Measuring acceptability of therapy (face validity). A self-reported measure of satisfaction regarding the content of the therapy. A questionnaire has been devised based on the theoretical framework of acceptability in Sekon, Cartwright & Francis (2017). There are two versions for post session one and post session eight with slightly different wording. This outcome measure will assess change.
Measure of adverse reactions | Participants will complete this before each therapy session weekly and it will be discussed with the therapist/PI in session. As therapy is for 8 weeks, participants will complete this once weekly for eight weeks.
  A quantitative measure containing a list of anticipated/likely adverse reactions (e.g. exacerbation of pain, feeling more upset than usual, increased problems in relationships) and unanticipated/adverse reactions. It is expected that therapy may increase emotional symptoms in the short term as the participants make realisations within therapy. This is a tick box measure with a qualitative 'other' box for further input.This outcome measure will assess change.
Objective measure of behaviour 2 - Completion rate from therapy | Measured at the end of therapy (at week 8).
  Measuring feasibility/acceptability of therapy

SECONDARY OUTCOMES:
Chronic Pain Acceptance Questionnaire-8 (CPAQ-8) | During baseline (no therapy) this will be completed weekly for a minimum of 3 weeks and a maximum of 6 weeks (dependent on randomised baseline group). All participants will complete the measure weekly during therapy for 8 weeks.
  CPAQ-8 - Fish, R. A., McGuire, B., Hogan, M., et al. (2010) A short version of the CPAQ and consists of eight items which measures pain acceptance and distress.
Pain Self Efficacy Questionnaire (PSEQ) | During baseline (no therapy) this will be completed weekly for a minimum of 3 weeks and a maximum of 6 weeks (dependent on randomised baseline group). All participants will complete the measure weekly during therapy for 8 weeks.
  PSEQ Nicholas, M. K (2007). The PSEQ assesses confidence in performing activities whilst in pain and beliefs about coping with pain.
The Interpersonal Needs Questionnaire for Pain (INQ-P) | During baseline (no therapy) this will be completed weekly for a minimum of 3 weeks and a maximum of 6 weeks (dependent on randomised baseline group). All participants will complete the measure weekly during therapy for 8 weeks.
  INQ-P (Methley et al. 2017). A measure of interpersonal factors in chronic pain adapted from the INQ; assesses thwarted belongingness and perceived burdensomeness specific to chronic pain.
The Beck Depression Inventory (BDI) | During baseline (no therapy) this will be completed weekly for a minimum of 3 weeks and a maximum of 6 weeks (dependent on randomised baseline group). All participants will complete the measure weekly during therapy for 8 weeks.
  BDI (Beck et al. 1961). The BDI is recommended as a core outcome measure of emotional functioning in chronic pain clinical trials (Dworkin at al., 2005).
Daily clinical measure (4 questions) | During baseline (no therapy) answered daily for a minimum of 3 weeks and a maximum of 6 weeks (dependent on randomised baseline group). All participants will answer them daily during therapy for 8 weeks.
  Four single item measures were generated using literature on interpersonal difficulties in chronic pain. All questions may be scored from 0-5; 0 being 'Not at all' and 5 being ' As good as I can feel/Extremely'.
  1. "How distressing has your pain been today?"
  2. "How lonely have you felt today?"
  3. "How good have you felt about your relationships with other people today?"
  4. "How good have you felt about yourself today?" Item 1 is based on generic numerical rating scales used to measure pain distress.
  Item 2 is a measure of social distress that we would expect to be amenable to change via PIT; it is an important outcome that overlaps with but is not the same as depression.
  Items 3 and 4 measure variables that PIT is designed to target and which we might expect to mediate any improvement in the other outcomes. Item 3 links with social connection (i.e., belongingness) and item 4 with perceived burdensomeness since how you feel about yourself influences whether you see yours.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Morgan, Principal Investigator — University of Manchester
Locations (1):
- The Walton Centre NHS Foundation Trust, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Participants will be required to consent to their anonymised outcome data (clinical measures and feasibility/acceptability measures) being used in similar research studies conducted at the University of Manchester.
Supporting Information: Study Protocol
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Requesters will be required to sign a data access agreement.